CLINICAL TRIAL: NCT07076147
Title: Breast Cancer Screening Adherence for Women at Moderate Risk for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-25-1; NCI-2025-04494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-25-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-07-07; First posted 2025-07-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete a questionnaire and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study assesses breast cancer screening adherence for women at moderately increased risk for developing breast cancer based on gene mutation status or empiric risk model estimates. It also seeks to determine facilitators and barriers to screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Among women without a history of breast cancer: to compare women with moderate risk breast cancer gene mutations (Mutation Carrier Group) to women with a 20-40% empiric lifetime risk of breast cancer (Empiric Risk Group) in terms of how likely they are to undergo recommended breast MRI screening.

OUTLINE: This is an observational study.

Patients complete a questionnaire and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * >= 30 years

  * =< 75 years
  * Women with either:

    * Genetic test results showing moderately increased breast cancer risk due to a pathogenic/likely pathogenic variant in ATM, CHEK2, BARD1, RAD51C, or RAD51D (Mutation carrier group) OR
    * Calculated lifetime breast cancer risk estimates between 20% and 40% according to the Tyrer-Cuzick V8.0B empiric risk model (Empiric risk group)
  * Patients provided breast cancer risk assessments by genetic counselors at USC Norris or LA General Hospital beginning in 2021 and at least 12 months ago
  * Women recommended to undergo annual breast MRI and/or annual mammogram beginning at the time of their genetic counseling risk assessment
  * English or Spanish speaking patients

Exclusion Criteria:

* * History of breast cancer before genetic counseling at University of Southern California (USC)

  * Any metastatic cancer diagnosis at time of genetic counseling risk assessment
  * Deceased
  * Patient underwent a risk reducing mastectomy before their genetic counseling risk assessment

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women provided with a breast cancer risk assessment by genetic counselors at USC Norris or LA General Hospital with either genetic test results showing moderately increased breast cancer risk due to a pathogenic/likely pathogenic variant in ATM, CHEK2, BARD1, RAD51C, or RAD51D or a calculated lifetime breast cancer risk estimates between 20% and 40% according to the Tyrer-Cuzick V8.0B empiric risk model who are recommended to undergo annual breast MRI and/or annual mammogram.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of women who undergo a screening breast MRI within 12 months of genetic test counseling | Up to 2 years
  Will be calculated for each of the 4 Hospital-by-Age subgroups for the 2 risk groups; then a one-sided, α=0.05 Mantel Haenszel test, stratifying by hospital and age, will be used to compare the Mutation Carrier Risk and the Empiric Risk groups in terms of adherence to screening MRI. Homogeneity of odds ratios will be tested to ensure that difference (odds ratio) between the two risk groups is fairly consistent across the 4 strata.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Comeaux, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California